CLINICAL TRIAL: NCT05648864
Title: Geographic Information System (GIS) Based Intervention 'Viamigo' for People With Dementia and Their Informal Caregivers: A Single-arm Trial to Evaluate the Feasibility and Preliminary Participant Responses
Brief Title: Viamigo for People With Dementia and Their Informal Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL81938.068.22
Record Dates: First submitted 2022-10-05; First posted 2022-12-13 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Dementia
Keywords: social participation; community; technology; mobile application; feasibility
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Masking Description: dyads of people living with dementia (n=24) and their informal caregivers (n=24)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Viamigo intervention (Experimental): All eligible and consenting dyads will be asked to participate in the Viamigo intervention (mobile application), consisting of three main components: (1) a face-to-face technology training session of 60 minutes, (2) a 3-month period of using the Viamigo intervention with support phone calls of approximately 5 minutes by the coordinating investigator once every two weeks, and (3) an evaluation phone call of 5-10 minutes.
  Interventions: Device: Viamigo

INTERVENTIONS:
Device: Viamigo — Mobile application with the aim to enhance the independent outdoor mobility of the user while a coach (informal caregiver) can monitor the route from a distance.

SUMMARY:
The main objective of this study is to evaluate the feasibility of the Geographic Information System (GIS)-based mobile application 'Viamigo' among people with dementia living in the community and their informal caregivers. Viamigo aims to support the independent out-of-home mobility of the user and to reduce informal caregiver's burden by teaching users a known individual route, which they can accomplish independently while being monitored by an informal caregiver. Although Viamigo was initially developed for persons with intellectual disabilities, it is expected that it can also support and improve out-of-home mobility and thereby the social participation of people with dementia. The design of the study is a mixed methods single-arm pre-post design with a baseline assessment, a 3-month intervention period, and a post-intervention assessment. Dyads (n=24) of people with mild to moderate dementia living in the community and their informal caregivers will use the mobile application for 3 months. The main study parameter is the feasibility of the Viamigo intervention for people with dementia and their informal caregivers. Secondary study parameters for people with dementia include out-of-home mobility and social participation. Secondary study parameters for informal caregivers include quality of life, caregiver burden, and gains in dementia caregiving.

DETAILED DESCRIPTION:
Rationale: People with dementia living in the community experience reduced out-of-home mobility and participate less in activities outside the home. This results in reduced social participation outside the home, which can negatively affect their health (e.g. leads to social isolation and increased risk of depressive symptoms). Technological interventions show promise in enhancing the social participation of people with dementia. However, there is a lack of technological interventions that facilitate social participation outside the home. While a growing body of evidence highlights the potential of Geographic Information Systems (GIS) in facilitating the out-of-home mobility of people with dementia and reducing informal caregivers' feelings of worry, very little attention is paid to the potential of GIS in enhancing the social participation of people with dementia. The GIS-based mobile application Viamigo aims to support the independent out-of-home mobility of the user and to reduce informal caregiver's burden by teaching users a known individual route, which they can accomplish independently afterwards while being monitored by an informal caregiver. Although Viamigo was initially developed for persons with intellectual disabilities, it is expected that it can also support and improve out-of-home mobility and thereby the social participation of people with dementia.

Objective: The main objective of this study is to evaluate the feasibility of the Viamigo intervention among people with dementia living in the community and their informal caregivers. The secondary objective of this study is to assess the first responses of people with dementia and informal caregivers to the Viamigo intervention.

Study design: This feasibility study includes a mixed methods single-arm pre-post design with a baseline assessment, a 3-month intervention period, and a post-intervention assessment.

Study population: The study population consists of dyads (n=24) of people with mild to moderate dementia living in the community and their informal caregivers. There are no restrictions regarding sex, educational level, or cultural background.

Intervention (if applicable): All eligible and consenting dyads will be asked to participate in the Viamigo intervention, consisting of three main components: (1) a face-to-face technology training session of 60 minutes, (2) a 3-month period of using the Viamigo intervention with support phone calls of approximately 5 minutes by the coordinating investigator once every two weeks, and (3) an evaluation phone call of 5-10 minutes.

Main study parameters/endpoints: The main study parameter is the feasibility of the Viamigo intervention for people with dementia and their informal caregivers. Secondary study parameters for people with dementia include out-of-home mobility and social participation. Secondary study parameters for informal caregivers include quality of life, caregiver burden, and gains in dementia caregiving.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: People with dementia will be asked to fill in the same two questionnaires (approximately 20 minutes in total) during the baseline and post-intervention assessment. Additionally, they are asked to fill in a daily travel diary for one week at baseline and during the last week of the intervention period. Informal caregivers will be asked to fill in the same three questionnaires (approximately 25 minutes in total) during the baseline and post-intervention assessment, and another 15-minutes questionnaire during the post-intervention assessment. Additionally, a smaller sample of the dyads (10 dyads) will be asked to share their experiences using the Viamigo intervention in a semi-structured post-intervention interview of approximately 30 minutes. Dyads will be asked whether they prefer to conduct the different assessments at home or at another location (e.g. Maastricht University). By participating in the study, a participant with dementia might be more often exposed to potentially risky situations in his or her living environment (e.g. traffic). Participation in a technological intervention study can be time-consuming and demanding. One way to reduce the burden of the study is to give participants the freedom to use the Viamigo application at their own pace.

ELIGIBILITY:
Inclusion Criteria people with dementia:

* Capacity to give informed consent;
* Diagnosis of mild to moderate dementia as evaluated by a healthcare professional and as reported by the person with dementia and the informal caregiver (by asking when and where the person has been diagnosed and by who);
* Living in the community (alone or with family/roommate(s)/friends);
* Taking part in social activities outside the home;
* Availability of an informal caregiver who is interested to take part in this study;
* Having an Android smartphone, as the Viamigo application to be used by the person with dementia is currently exclusively available for Android.

Inclusion criteria informal caregivers:

* Family caregiver of participant diagnosed with mild to moderate dementia;
* Aged 18+;
* Having at least weekly contact with the person with dementia;
* Having an Android or Apple smartphone and laptop/computer.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* No informed consent given;
* Concurrent participation in any other interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Overall feasibility of Viamigo intervention | 3 months
  Semi-structured interviews with dyads (participants with dementia and informal caregivers)
Recruitment and drop-out rates | 3 months
  Number of referred dyads, number of eligible participants who are willing to participate, number of eligible participants who are not willing to participate, including reasons for declined participation (if provided); number of dropouts during the baseline assessment (after signing informed consent and before starting the intervention) as well as reasons for dropout, if provided; number of dropouts after starting the intervention and reasons for dropout, if provided
Recruitment time | 3 months
  Amount of spent time on recruiting participants (recruitment capability) in weeks
Data collection methods of Viamigo intervention | 3 months
  Notes on: if outcome measures were sensitive to change; how understandable data collection procedures were for study participants; and how much time was required to fill in questionnaires
Social validity of Viamigo intervention | 3 months
  measured by selfreported Program Participation Questionnaire (PPQ)
Practicality of Viamigo intervention | 3 months
  Practical constraints in the context and environment to implement the Viamigo intervention (e.g.
  time or resource availability) will be tracked with notes
Adaptability of Viamigo intervention | 3 months
  Aspects facilitating or impeding the flexibility of the intervention, as well as a potential needed set of requirements to implement the intervention with people with dementia and their informal caregivers will be tracked with notes

SECONDARY OUTCOMES:
Change in out-of-home mobility of participants with dementia at 3 months | 3 months
  Measured by a travel diary
Change in social participation of participants with dementia at 3 months | 3 months
  Measured by the Engagement and Independence in Dementia Questionnaire (EID-Q), the Lubben Social Network Scale - 6 (LSNS-6), and the post-intervention semi-structured interview
Change in quality of life of informal caregivers at 3 months | 3 months
  Measured by the Investigating Choice Experiments CAPability measure for Older people (ICECAP-O)
Change in caregiver burden at 3 months | 3 months
  Measured by the Burden Scale for Family Caregivers - short version (BSFC-s)
Change in gains in dementia caregiving at 3 months | 3 months
  Measured by Gain in Alzheimer care INstrument (GAIN)

OTHER OUTCOMES:
Stage of dementia | week 0 (baseline)
  Measured by the Clinical Dementia Rating (CDR)

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein E. de Vugt, Prof., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, an anonymised version of the data will be made available for reuse on a data repository, such as Dataverse.nl. No personal data will be included. Access to this data will be allowed under specified conditions (still in discussion with the legal advisor of Maastricht University). All participants will be asked for consent to reuse their data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymised data will become available right after the completion of the study. All data will be securely stored and available for 15 years after the last publication on the data.
Access Criteria: Access to the data collection will be restricted by conditions for use. These conditions will be determined in consultation with a legal adviser of Maastricht University. The legal adviser has been contacted via e-mail (privacy@maastrichtuniversity.nl).